CLINICAL TRIAL: NCT07183943
Title: Visual Reality Gaming Based Proprioceptive Neuromuscular Facilitation on Spatiotemporal Parameters in Upper Limb Burned Patients
Brief Title: VR Gaming Based PNF on Spatiotemporal Parameters in Upper Limb Burned Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: MTI University (Other)
Responsible Party: Principal Investigator, Ahmed Mohamed Ahmed Abd El hady El Fahl,ph.d, Assisstant professor, MTI University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P.T.REC/012/005914
Record Dates: First submitted 2025-09-08; First posted 2025-09-19 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Burns
MeSH Terms: conditions — Burns | interventions — Muscle Stretching Exercises

STUDY DESIGN:
Intervention Model Description: RCT
Who Masked: Participant, Outcomes Assessor
Masking Description: Double blinded
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Proprioceptive neuromuscular facilitation (PNF) (Experimental): In the PNF group, The PNF sequence included scapula, upper limb, Training was performed in different positions
  Interventions: Other: Proprioceptive neuromuscular facilitation (PNF)
- Visual reality (VR) (Experimental): In the VR group, the tasks were performed with the aid of a Nintendo Wii device.
  Interventions: Other: Visual reality (VR)
- PNF and VR (Experimental): The PNF/VR group performed both PNF and VR exercises. The duration of the exercises was modified so that half of the time was devoted to PNF and the other half to VR
  Interventions: Other: PNF and VR
- Control group (No Intervention): No intervention

INTERVENTIONS:
Other: Proprioceptive neuromuscular facilitation (PNF) — Training was performed in different positions (decubitus, sitting, and standing) according to the specific exercise. the participants performed 10 minutes of diagonal scapula exercises (anterior and posterior elevation) and 30 minutes of upper limb diagonals (Flexion-Abduction-External Rotation and Extension-Abduction-Internal Rotation), including the 5 initial minutes of stretching.
  Arms: Proprioceptive neuromuscular facilitation (PNF)
Other: Visual reality (VR) — The site of the intervention was a 20-square-meter room equipped with a multimedia projector, which projected the image on the wall at a height of 1 m and 20 cm. A professional physical therapist supervised the treatment continuously, and every participant received prior instructions on the conduct of the games. The therapeutic protocol included 4 electronic games: Balance Bubble Plus, Rhythm Parade, Tennis, and Box.
  Arms: Visual reality (VR)
Other: PNF and VR — The total duration of the sessions remained consistent. The participants performed 5 minutes of scapula diagonals and 15 minutes of upper limb diagonals in the weekly session. The games for the PNF/VR group were the same as those for the VR group, except for their duration. Whereas they were performed for 20 minutes each in the VR group, the session including 5 minutes of stretching.
  Arms: PNF and VR

SUMMARY:
Burn injuries are among the most severe forms of trauma, often leading to significant physical and psychological challenges. The rehabilitation process for burn patients, particularly those with upper limb injuries, is complex due to the need for restoring functional movement and reducing scar contracture. Traditional rehabilitation methods focus on restoring range of motion, muscle strength, and coordination. However, these approaches can be limited in engaging patients and maintaining their motivation throughout the recovery process.

DETAILED DESCRIPTION:
Upper limb burn injury (ULBI) often leads to significant dysfunction . Severe pain, limited range of motion in the joint and kinesiophobia may affect upper limb functionality and activities of daily living in the acute term of injury . Increased pain and limitations in range of motion and function of the upper limb may cause deterioration in reciprocal arm swing which plays a substantial role in gait pattern by contributing to the co-ordination of the trunk, pelvis and leg movements, reducing energy expenditure and improving gait stability and balance.

Proprioceptive Neuromuscular Facilitation (PNF) is a therapeutic exercise technique used to enhance both passive and active range of motion with the aim of improving neuromuscular control and coordination. By integrating PNF with innovative technologies such as Virtual Reality (VR) gaming systems, rehabilitation can be transformed into an engaging and immersive experience. VR provides a unique environment that can simulate real-life scenarios, offering a controlled yet dynamic setting that encourages active participation and motivation.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of unilateral upper extremity burn injury
* must be able to walk independently
* Agreeing to participate voluntarily in the study
* 18-65 years of age
* the ability to accurately express the level of pain that prevents cognitive, affective and verbal communication

Exclusion Criteria:

* Walking with assist device
* Having a visual deficits
* Having an orthopedic problems that affect gait
* Having a neurological disorders
* Having a musculoskeletal disorders that affect gait
* Having an undergone orthopedic surgery

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2025-10-01 (Actual); Primary Completion 2026-01-01 (Actual); Study Completion 2026-01-05 (Actual)

PRIMARY OUTCOMES:
Kinesiophobia | at baseline and at 12 weeks
  the Arabic version of the Tampa Scale for Kinesiophobia (TSK) was used. The TSK is rated on a 4-point Likert scale ranging from 17 to 68, with higher scores indicating a high level of kinesiophobia . The TSK has been shown to be a reliable tool for the measurement of kinesiophobia in patients with (upper limb burn injury) ULBI.

SECONDARY OUTCOMES:
Gait Analysis | at baseline and at 12 weeks
  The GAITRite (CIR System INC. Clifton, NJ, USA, 07012) electronic walkway was used to evaluate the spatio-temporal parameters during walking. Participants walked barefoot at self-selected pace. Gait analysis was started after a trial to allow the participants to become familiar with the test. Gait velocity, cadence and bilateral gait parameters of step length, stride length, percentage of stance and swing were used for analysis. In addition spatio-temporal parameters and plantar pressure distribution were analyzed during walking. The GAITRite system expresses the plantar pressure value as a percentage of the maximum pressure.
Arm swing | at baseline and at 12 weeks
  The arm swing movements during walking were evaluated with free version of Kinovea 2D motion analysis software (Kinovea 0.8.15., GPLv2 license, 2019). It is a reliable method to analyze the upper extremity movements and gait analysis . For tracking the segments of the upper limbs during walking, sticker markers were placed in specific anatomical areas (left/right acromions, left/right medial and lateral epicondyles, and left/right distal radius and ulna landmarks) . The shoulder, elbow, and wrist joints were manually positioned within the Kinovea software to accurately map the participants' upper body movements. Based on the identified joint centers, the upper arm, lower arm, and full arm segments were determined. Detailed analyses were conducted to evaluate the shoulder angle (measured from the shoulder joint marker to the elbow joint marker), the elbow angle (measured from the elbow joint marker to the midpoint of the wrist joint marker).

CONTACTS AND LOCATIONS:
Locations (1):
- faculty of physical therapy ,Cairo University, Cairo, Egypt